CLINICAL TRIAL: NCT02239380
Title: A Multi-center, Open-label, Non-controlled Study To Evaluate The Efficacy And Safety Of Lorazepam Intravenously Administered In Subjects With Status Epilepticus Or Repetitive Status Epilepticus
Brief Title: Lorazepam for the Treatment of Status Epilepticus or Repetitive Status Epilepticus in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B3541002; 2017-000125-13 (EudraCT Number)
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2018-10

CONDITIONS: Status Epilepticus
Keywords: Lorazepam; Status Epilepticus
MeSH Terms: conditions — Status Epilepticus | interventions — Lorazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lorazepam (Experimental): Lorazepam intravenous formulation
  Interventions: Drug: Lorazepam

INTERVENTIONS:
Drug: Lorazepam — intravenous administration. Dosage for adult subjects (16 years aged and over): 4 mg Dosage for pediatric subjects (3 months to < 16 years): 0.05 mg/kg (but not exceeding 4 mg) Frequency: Intravenous administration of lorazepam. Subjects whose seizure does not stop or recurs within 10 minutes after the initial dose may receive the same amount of lorazepam injection no earlier than 10 minutes following the initial dose.
  Also, subjects whose seizure stops within 10 minutes after the initial dose, but recurs thereafter (within 12 hours) may receive the same amount of lorazepam injection; a total of 2 doses will be permitted in this study.

SUMMARY:
The purpose of this study is to determine the efficacy, safety and pharmacokinetics of Lorazepam on Japanese patients with Status Epilepticus or Repetitive Status Eplilepticus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with status epilepticus or repetitive status epilepticus / cluster seizure who have seizures that can be evaluated by investigator's visual observations based on motor symptoms or who have seizures that can be evaluated by EEG.
* Subjects with status epilepticus accompanied by generalized seizure, partial seizure or secondarily generalized seizure lasting 5 minutes or longer
* Subjects with repetitive status epilepticus / cluster seizure accompanied by not less than 3 consecutive episodes of generalized seizure, partial seizure or secondarily generalized seizure in 1 hour.
* Subjects not younger than 3 months (either gender is eligible for the study)

Exclusion Criteria:

* Subjects with known or suspected recurrent seizures due to illegal drug or alcohol withdrawal
* Subjects with known history of hypersensitivity to lorazepam or benzodiazepine
* Subjects with a known history of benzodiazepine abuse.
* Subjects currently receiving lorazepam
* Subjects with angle-closure glaucoma
* Subjects with myasthenia gravis
* Subjects with either of aspartate transaminase, alanine transaminase, total bilirubin, blood urea nitrogen, or creatinine at screening visit exceeding 2x the upper limit of normal of the institutional reference value (if the data is available)
* Subjects with white blood cell count less than 3000/mm3 or neutrophil count less than 1500/mm3 at screening visit (if the data is available)

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (20):
- Japan (20):
  - Aichi Children's Health and Medical Center, Obu-shi, Aichi-ken
  - National Hospital Organization Fukuoka-Higashi Medical Center, Koga, Fukuoka
  - Hokkaido Medical Center for Child Health and Rehabilitation, Sapporo, Hokkaido
  - Nakamura Memorial Hospital, Sapporo, Hokkaido
  - National Hospital Organization Hokkaido Medical Center, Sapporo, Hokkaido
  - Hyogo Prefectural Kobe Children's Hospital, Kobe, Hyōgo
  - Tohoku University Hospital, Sendai, Miyagi
  - National Hospital Organization Nagasaki Medical Center, Ohmura, Nagasaki
  - National Nishi-Niigata Central Hospital / Pediatrics, Niigata, Niigata
  - Okayama University Hospital / Child Neurology, Okayama, Okayama-ken
  - Osaka Medical Center and Research Institute for Maternal and Child Health, Izumi, Osaka
  - Osaka City General Hospital Pediatric Neurology, Miyakojima-ku, Osaka
  - NHO Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka, Shizuoka
  - National Center of Neurology and Psychiatry, Kodaira, Tokyo
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi
  - Fukuoka Children's Hospital, Fukuoka
  - Fukuoka Sanno Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Gifu Prefectural General Medical Center, Gifu
  - Saitama Children's Medical Center, Saitama

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3541002&StudyName=Lorazepam%20for%20the%20Treatment%20of%20Status%20Epilepticus%20or%20Repetitive%20Status%20Epilepticus%20in%20Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Lorazepam: Participants aged between 3 months to below 16 years received single intravenous dose (Dose 1) of 0.05 milligram per kilogram (mg/kg) of Lorazepam (up to a maximum dose of 4 mg) on Day 1. Participants aged above 16 years received single intravenous dose of 4 mg of Lorazepam. Participants whose seizures continued or recurred within 10 minutes following the initial dose, an additional dose (Dose 2) of 4 mg (for participants above 16 years of age) or 0.05 mg/kg dose (for participants between 3 months to below 16 years of age) was administered accordingly. Participants were followed up to 7 days after last dose of study drug administration.
Period: Overall Study
Arm/Group | Lorazepam
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Arm/Group | Lorazepam
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.0 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Seizure Free Interval of At Least 30 Minutes After Initial Dose (Dose 1) of Study Drug
Description: Participants with clinical benefit were defined as participants whose initial seizure stopped within 10 minutes after initial dose (Dose 1) and who continued seizure-free for at least 30 minutes after the completion of initial dose (Dose 1).
Time Frame: 30 minutes post Dose 1
Population: Full analysis set (FAS) included all participants who received at least 1 dose of study drug, excluded those participants whose status epilepticus (SE) or repetitive SE/cluster seizure was determined on the electroencephalography (EEG).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lorazepam
Number analyzed (Participants) | 25
percentage of participants | 48.0 [27.8 to 68.7]

2. Secondary Outcome: Percentage of Participants Who Achieved Seizure Free Interval of At Least 30 Minutes After Any Dose of Study Drug
Description: Percentage of participants whose initial seizure stopped within 10 minutes after the administration of study drug (either Dose 1 or 2 [in 10 to 30 minutes from the initial dose]) and who continued seizure-free for at least 30 minutes were analyzed and reported in this outcome measure.
Time Frame: 30 minutes post Dose 1 or 2
Population: FAS included all participants who received at least 1 dose of study drug, excluded those participants whose SE or repetitive SE/cluster seizure was determined on the EEG.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Lorazepam
Number analyzed (Participants) | 25
percentage of participants | 64.0 [42.5 to 82.0]

3. Secondary Outcome: Percentage of Participants Who Achieved Seizure Free Interval of At Least 12 Hours After Administration (Either Initial or Any Dose) of Study Drug
Description: Percentage of participants whose seizures stopped within 10 minutes after the administration of initial dose (Dose 1) of study drug and after any study drug dose (either Dose 1 or Dose 2 [in 10 to 30 minutes from the initial dose]), who continued to be seizure-free for at least 12 hours post-dose were analyzed and reported in this outcome measure.
Time Frame: 12 hour post Dose 1; 12 hour post Dose 1 or 2
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Lorazepam
Number analyzed (Participants) | 25
percentage of participants
  Post Dose 1 | 32.0
  Post Dose 1 or 2 | 44.0

4. Secondary Outcome: Percentage of Participants Who Achieved Seizure Free Interval of At Least 24 Hours After Administration (Either Initial or Any Dose) of Study Drug
Description: Percentage of participants whose seizures stopped within 10 minutes after the administration of initial dose (Dose 1) of study drug and after any study drug dose (either Dose 1 or Dose 2 [in 10 to 30 minutes from the initial dose]), who continued to be seizure-free for at least 24 hours post-dose were analyzed and reported in this outcome measure.
Time Frame: 24 hour post Dose 1; 24 hour post Dose 1 or 2
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Lorazepam
Number analyzed (Participants) | 25
percentage of participants
  Post Dose 1 | 24.0
  Post Dose 1 or 2 | 32.0

5. Secondary Outcome: Time to Resolution of Seizures From The Administration (Either Initial or Any Dose) of Study Drug
Description: Time to resolution (in minutes) was defined as the duration between the administration of study drug until the seizure resolved without receiving the prohibited medications.
Time Frame: 10 minutes post Dose 1; 10 minutes post Dose 1 or 2
Population: FAS included all participants who received at least 1 dose of study drug, excluded those participants whose SE or repetitive SE/cluster seizure was determined on the EEG. Here, 'n' signifies those participants who were evaluable for specific category.
Measure: Median (Full Range); unit: minutes
Arm/Group | Lorazepam
Number analyzed (Participants) | 25
minutes
  Post Dose 1: number analyzed (Participants) | 15
  Post Dose 1 | 1.0 [0 to 10]
  Post Dose 1 or 2: number analyzed (Participants) | 17
  Post Dose 1 or 2 | 1.0 [0 to 10]

6. Secondary Outcome: Time to Relapse Following The Administration (Either Initial or Any Dose) of Study Drug
Description: Time to relapse (in minutes) was defined as duration from the time of study drug administration to the time of relapse, as determined by investigator. Participants whose seizure stops within 10 minutes without receiving the prohibited medications were analyzed in this outcome measure.
Time Frame: 24 hour post Dose 1; 24 hour post Dose 1 or 2
Population: FAS included all participants who received at least 1 dose of study drug, excluded those participants whose SE or repetitive SE/cluster seizure was determined on the EEG. Here, number of participants analyzed (N) signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: minutes
Arm/Group | Lorazepam
Number analyzed (Participants) | 9
minutes
  Post Dose 1 | 62.0 [11 to 879]
  Post Dose 1 or 2 | 103.0 [23 to 1246]

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug to the end of study (Day 12), that were absent before treatment or that worsened relative to pre-treatment state. AEs include both serious and non-serious adverse events.
Time Frame: Baseline up to 7 days after last dose of study drug administration (up to 12 days)
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Lorazepam
Number analyzed (Participants) | 26
participants
  AEs | 12
  SAEs | 1

ADVERSE EVENTS:
Time Frame: Baseline up to 7 days after last dose of study drug administration (up to 12 days)
Description: The same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in one event and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Lorazepam
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 12/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lorazepam (N=26)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lorazepam (N=26)
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Ataxia (Nervous system disorders) | 1
Balance disorder (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 2
Pollakiuria (Renal and urinary disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.